CLINICAL TRIAL: NCT02845908
Title: A Phase 2 Study of POF(Paclitaxel/Oxaliplatin/5-Fluorouracil/Leucovorin) Versus FOLFOX Versus FOLFOX Plus Intraperitoneal Paclitaxel as a First-line Treatment in Advanced Gastric Cancer
Brief Title: POF Versus FOLFOX Versus FOLFOX Plus ip Paclitaxel in AGC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF-004
Record Dates: First submitted 2016-06-28; First posted 2016-07-27 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-03

CONDITIONS: Malignant Neoplasm of Stomach Stage IV
MeSH Terms: conditions — Stomach Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- POF (Experimental): The POF regimen consisted of a 3-hour infusion of paclitaxel (135 mg/m2) followed by oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days. The combined chemotheraphy will be treated for 9 circle. then，the capetabine was allowed
  Interventions: Drug: POF; Drug: FOLFOX; Drug: FOLFOX plus PAC(ip)
- FOLFOX plus PAC(ip) (Experimental): The regimen consisted of oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2) plus paclitaxel (80 mg/m2) intra-peritoneally.Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.
  Interventions: Drug: POF; Drug: FOLFOX; Drug: FOLFOX plus PAC(ip)
- FOLFOX (Active Comparator): The FOLFOX regimen consisted of oxaliplatin (85 mg/m2) and Calcium Levofolinate (200 mg/m2).Subsequently, a 46-hour infusion of fluorouracil (2400 mg/m2) was administered using an ambulatory pump, repeating the cycle every 14 days.
  Interventions: Drug: FOLFOX; Drug: FOLFOX plus PAC(ip)

INTERVENTIONS:
Drug: POF — Paclitaxel plus Oxaliplatin plus Leucovorin plus 5-FU
  Arms: FOLFOX plus PAC(ip); POF
Drug: FOLFOX — Oxaliplatin plus Leucovorin plus 5-FU
Drug: FOLFOX plus PAC(ip) — FOLFOX plus intraperitoneally PAC

SUMMARY:
The aim of this study was to compare the efficacy and safety of POF, FOLFOX, and FOLFOX plus paclitaxel(ip) as first-line treatment in AGC a phase II clinical trial.

DETAILED DESCRIPTION:
The biweekly 5-fluorouracil and leucovorin (LV5FU2) regimen associated with oxaliplatin (FOLFOX) is active in patients with AGC. Meanwhile, Paclitaxel monotherapy is also active in patients with AGC. In previous studies, we found that POF(A combination of oxaliplatin, fluorouracil and Paclitaxel) regimen appears to be of good efficacy and is well tolerated in patients with advanced gastric cancer. This study is being done to find out if three drugs combination maintain manageable side effects but have better benefit than two drugs combination. Intraperitoneal paclitaxel showed high local concentration in abdominal cavity and low systemic toxicity. This study is being done to find out if the combination with Intraperitoneal paclitaxel and FOLFOX have higher local control rate and lower systemic toxicity.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-75 years;
2. Patients must have histologically or cytologically confirmed metastatic or unresectable gastric or gastroesophageal junction (GEJ) adenocarcinoma. GEJ adenocarcinoma may be classified according to Siewert's classification type I, II, or III. Histological documentation of local recurrence or metastasis is strongly encouraged, unless the risk of such a procedure outweighs the potential benefit of confirming the metastatic disease;
3. Patients must have disease that can be measurable radiographically measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1);
4. Patients may have received no prior chemotherapy for metastatic or unresectable disease. Patients may have received prior adjuvant therapy (chemotherapy and/or chemoradiation) if more than 6 months have elapsed between the end of adjuvant therapy and registration.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1;
6. An expected survival of ≥3months;
7. Major organ function has to meet the following criteria: (1) For results of blood routine test: Hemoglobin (HB) ≥80 g/L, ANC (absolute neutrophil count) ≥1.5 × 109/L, PLT (blood platelet) ≥75 × 109/L; (2) For results of biochemical tests: BLT (total bilirubin) ≤1.25 × the upper limit of normal (ULN), ALT (Alanine aminotransferase) and AST (aspartate aminotransferase ) ≤2.5 × ULN, liver metastases, if any, the ALT and AST ≤5 × ULN, Serum Cr（creatinine）≤1 × ULN, Endogenous creatinine clearance rate >50ml/min;
8. The patient has an INR (international normalized ratio) ≤1.5 and an PTT（Partial Thromboplastin Time）≤3 seconds above the ULN if the patient is not on anticoagulation. If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment: (1) The patient must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of LMW (Low molecular weight) heparin; (2) The patient must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices)
9. Pregnancy test (serum or urine) has to be performed for woman of childbearing age within 7 days before enrolment and the test result must be negative. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
10. Ability to understand informed consent and signing of written informed consent document prior to initiation of protocol therapy.

Exclusion criteria:

1. Patients who have ascites requiring frequent drainage;
2. Patients who have received previous chemotherapy for the treatment of metastatic or unresectable gastric or GEJ adenocarcinoma are ineligible;
3. Patients who have received previous pre- or post-operative chemotherapy or chemoradiation are ineligible if therapy was completed less than 6 months prior to study registration;
4. Patients with a history of another neoplastic disease within the past three years, excluding basal cell carcinoma of the skin, cervical carcinoma in situ, or nonmetastatic prostate cancer;
5. Patients with brain or central nervous system metastases, including leptomeningeal disease;
6. Pregnant (positive pregnancy test) or breast feeding;
7. Serious, non-healing wound, ulcer, or bone fracture;
8. Significant cardiac disease as defined as: unstable angina, New York Heart Association (NYHA) grade II or greater, congestive heart failure, history of myocardial infarction within 6 months;
9. Evidence of bleeding diathesis or coagulopathy;
10. History of a stroke or CVA within 6 months;
11. Clinically significant peripheral vascular disease;
12. Peripheral neuropathy grade ≥2 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03;
13. Inability to comply with study and/or follow-up procedures;
14. Patients with any other medical condition or reason, in that investigator's opinion, makes the patient unstable to participate in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival,PFS | 9 month
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival).

SECONDARY OUTCOMES:
Response Rate, RR | 9 month
  Response rate per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Adverse Event（AE） | 6month
  Clinical response of treatment according to RESIST v1.1 criteria (ORR, According to NCI CTCAE 4.03 criteria
The EORTC Core Quality of Life questionnaire (QLQ-C30): | 6month
  a quality-of-life instrument for use in international clinical trials in oncology.
EORTC quality of life questionnaire to assess chemotherapy-induced peripheral neuropathy,QLQ-CIPN20 | 6 month
  EORTC quality of life questionnaire to assess chemotherapy-induced peripheral neuropathy
Overall Survival(OS) | 12 months
  The length of time from enrollment until the time of death (OS, overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Rongbo Lin, MD, Study Chair — Fujian Cancer Hospital
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China